CLINICAL TRIAL: NCT06464367
Title: Mechanistic Studies of Psilocybin in Headache Disorders
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Wallace Foundation (Other)
Responsible Party: Principal Investigator, Emmanuelle Schindler, Assistant Professor of Neurology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000034634; ES0006 (Other: VA Connecticut Healthcare System)
Record Dates: First submitted 2024-06-08; First posted 2024-06-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Migraine
Keywords: psilocybin; resting state functional connectivity; synaptic density; synaptic vessel glycoprotein 2A (SV2A); circadian rhythm; sleep; inflammation
MeSH Terms: conditions — Migraine Disorders; Inflammation | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Migraine psilocybin (Experimental): Migraine participants randomized to receive 10 mg psilocybin (oral)
  Interventions: Drug: Psilocybin
- Migraine placebo (Placebo Comparator): Migraine participants randomized to receive 2.5 mg THC (oral)
  Interventions: Drug: Placebo
- Healthy control psilocybin (Experimental): Healthy control participants randomized to receive 10 mg psilocybin (oral)
  Interventions: Drug: Psilocybin
- Healthy control placebo (Placebo Comparator): Healthy control participants randomized to receive 2.5 mg THC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — synthetic psilocybin 10 mg (oral)
  Arms: Healthy control psilocybin; Migraine psilocybin
Drug: Placebo — synthetic THC 2.5 mg (oral)
  Arms: Healthy control placebo; Migraine placebo

SUMMARY:
In previous clinical trial work, the investigators observed lasting reductions in headache burden after limited dosing of psilocybin. This purpose of this study is to examine potential sources for this observed effect. This study will measure brain resting state functional connectivity (fMRI), central synaptic density (SV2A PET), peripheral markers of inflammation, circadian rhythm (actigraphy), and sleep (sleep EEG) in both migraine and healthy control participants before and one week after the administration of psilocybin or an active control agent.

ELIGIBILITY:
Inclusion criteria:

* Age 21 to 70 (inclusive)
* Migraine disease per ICHD-3 criteria (for migraine participants) OR Healthy control patient

Exclusion criterion

* Unstable medical condition or serious nervous system pathology
* Pregnant, breastfeeding, lack of adequate birth control
* Psychotic or manic disorder
* Substance abuse in the prior 3 months
* Use of classic psychedelics (e.g., psilocybin, LSD, mescaline) in the past 6 months
* Use of cannabis or other THC products in the prior 2 weeks
* Urine toxicology positive to drugs of abuse
* The use of triptans (e.g., sumatriptan) or ditans (e.g., lasmiditan) more than twice weekly on average
* Use of serotonergic preventive therapies (i.e., taken chronically; amitriptyline, fluoxetine, imipramine, cyproheptadine) in the past 6 weeks
* Use of preventive or transitional treatments that produce spikes and waning of symptom relief (e.g., botulinum toxin, calcitonin gene-related peptide system targeting antibodies, peripheral nerve or ganglion blocks, chiropractic manipulation)
* History of a bleeding disorder or are currently taking anticoagulants (e.g., warfarin, enoxaparin, dabigatran, apixaban).
* Use of non-steroidal anti-inflammatory drugs (NSAIDs; e.g., ibuprofen, naproxen) in the 7 days before PET scan and 7 days after PET scan.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline SV2A PET | from date of randomization until the date of first PET scan, assessed up to 6 months
  Comparing initial SV2A PET between migraine and HC
Baseline RSFC | from date of randomization until the date of first MRI, assessed up to 6 months
  Comparing initial RSFC between migraine and HC
Change in SV2A PET after drug administration | from date of first PET scan to the date of second PET scan, assessed up to 6 months
  Comparing change in SV2A PET after drug between psilocybin/THC and migraine/HC
Change in resting state functional connectivity (RSFC) after drug administration | from date of first MRI to the date of second MRI, assessed up to 6 months
  Comparing change in RSFC after drug between psilocybin/THC and migraine/HC

SECONDARY OUTCOMES:
Change in TNF-alpha | from screening to 7 days after drug administration
  Comparing change in TNF-alpha levels after drug between psilocybin/THC and migraine/HC
Change in IL-1beta | from screening to 7 days after drug administration
  Comparing change in IL-1beta levels after drug between psilocybin/THC and migraine/HC
Change in IL-6 | from screening to 7 days after drug administration
  Comparing change in IL-6 levels after drug between psilocybin/THC and migraine/HC
Change in calcitonin gene-related peptide (CGRP) | from screening to 7 days after drug administration
  Comparing change in CGRP levels after drug between psilocybin/THC and migraine/HC
Change in pituitary adenylate cyclase activating polypeptide (PACAP) | from screening to 7 days after drug administration
  Comparing change in PACAP levels after drug between psilocybin/THC and migraine/HC
Change in bedtime (via actigraphy) | from screening through 14 days after drug administration
  Comparing change in bedtime (time) after drug between psilocybin/THC and migraine/HC
Change in get-up time (via actigraphy) | from screening through 14 days after drug administration
  Comparing change in get-up time (time) after drug between psilocybin/THC and migraine/HC
Change in daily active period (via actigraphy) | from screening through 14 days after drug administration
  Comparing change in daily active period (hours) after drug between psilocybin/THC and migraine/HC
Change in daily rest period (via actigraphy) | from screening through 14 days after drug administration
  Comparing change in daily rest period (hours) after drug between psilocybin/THC and migraine/HC
Change in REM latency (via sleep electroencephalography) | from screening to 7 days after drug administration
  Comparing change in REM latency (minutes) after drug between psilocybin/THC and migraine/HC
Change in percent REM (via sleep electroencephalography) | from screening to 7 days after drug administration
  Comparing change in percent REM (%) after drug between psilocybin/THC and migraine/HC
Change in sleep efficiency (via sleep electroencephalography) | from screening to 7 days after drug administration
  Comparing change in sleep efficiency (%) after drug between psilocybin/THC and migraine/HC
Adverse events | from screening through 3 months after drug administration
  Adverse events from any procedure or drug administration

OTHER OUTCOMES:
Acute change in TNF-alpha during drug administration | 0, 120, and 240 minutes after drug administration
  Comparing change in TNF-alpha between psilocybin/THC and migraine/HC
Acute change in IL-1beta during drug administration | 0, 120, and 240 minutes after drug administration
  Comparing change in IL-1beta between psilocybin/THC and migraine/HC
Acute change in IL-6 during drug administration | 0, 120, and 240 minutes after drug administration
  Comparing change in IL-6 between psilocybin/THC and migraine/HC
Acute change in calcitonin gene related peptide (CGRP) during drug administration | 0, 120, and 240 minutes after drug administration
  Comparing change in CGRP between psilocybin/THC and migraine/HC
Acute change in pituitary adenylate cyclase activating polypeptide (PACAP) during drug administration | 0, 120, and 240 minutes after drug administration
  Comparing change in PACAP between psilocybin/THC and migraine/HC
Acute change in mean arterial pressure (MAP) during drug administration | 0, 30, 60, 120, 180, 240, 300, and 360 minutes after drug administration
  Comparing change in MAP (mmHg) between psilocybin/THC and migraine/HC
Acute change in heart rate during drug administration | 0, 30, 60, 120, 180, 240, 300, and 360 minutes after drug administration
  Comparing change in heart rate (beats per minute) between psilocybin/THC and migraine/HC
Acute change in SpO2 during drug administration | 0, 30, 60, 120, 180, 240, 300, and 360 minutes after drug administration
  Comparing change in SpO2 (%) between psilocybin/THC and migraine/HC
Acute change in general drug effects during drug administration | 0, 30, 60, 120, 180, 240, 300, and 360 minutes after drug administration
  Comparing "overall," "anxiety/fear," "sleepiness/sedation," "nausea," "joy/intense happiness,""peace/harmony" between psilocybin/THC and migraine/HC
Acute psychedelic effects during drug administration | up to 8 hours after drug administration
  Comparing 5-Dimensional Altered States of Consciousness scale scores (0-100; higher score being more psychedelic) between psilocybin/THC and migraine/HC

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States